CLINICAL TRIAL: NCT06845657
Title: Effect of Hip Abductor Strengthening Exercises in Patients With Knee Osteoarthritis
Brief Title: Hip Abductor Strengthening Exercises in Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fouzia Kousar
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis
Keywords: Hip Abductor Strengthening; Muscle weakness; knee pain
MeSH Terms: conditions — Osteoarthritis, Knee; Muscle Weakness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip Abductor Strengthening Exercises+ Conventional PT (Active Comparator)
  Interventions: Other: Hip Abductor Strengthening Exercises
- Conventional PT (Other)
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Other: Hip Abductor Strengthening Exercises — Hip Abductor Strengthening Exercises .1.side lying leg raise 2.clam shell(Frequency: 3 sets 10 reps in session 1-5) 3.standing hip abduction.4.pelvic lift training (Frequency: 3 sets 10 reps in session 6-9) .Conventional PT including 1-ROM 2- Stretching of hamstrings,calf,,rectus femoris (30 sec hold,15 sec relaxation period,3 rep) 3.knee isometrics (2 sets 10 rep in first 5 sessions and 3 sets 10 rep in next 4 sessions).total duration is 3 sessions per week for 3 consecutive weeks.
  Arms: Hip Abductor Strengthening Exercises+ Conventional PT
Other: Conventional Treatment — Conventional PT including 1-ROM 2- Stretching of hamstrings,calf,rectus femoris (30 sec hold,15 sec relaxation period,3 rep) 3.knee isometrics (2 sets 10 rep in first 5 sessions and 3 sets 10 rep in next 4 sessions). Total duration is 3 sessions per week for 3 consecutive weeks
  Arms: Conventional PT

SUMMARY:
The aim of this randomized controlled trial is to find the effect of hip abductor strengthening exercises on pain, range of motion, functional disability and balance in patient with knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a chronic disease affecting the joint and its tissues, primarily leading to progressive damage to articular cartilage and, subsequently, to the subchondral bone and surrounding synovial structures. This chronic degenerative disease affects approximately one-third of adults, and its prevalence increasing with advancing age. The knee is one of the most common joints affected by the OA. Systematic reviews indicate a global prevalence of knee osteoarthritis (KOA) is 22.9% among individuals aged 40 and older, affecting an estimated 654.1 million people worldwide, with variations across countries and increasing with age.

Knee osteoarthritis (KOA) is a multi etiological, chronic disabling disease that affects the entire knee joint, which is the most common site of involvement in OA. KOA patients mostly suffer from progressive stiffness and knee pain. Gradually, they have some difficulties in performing daily activities, such as walking, squatting, and climbing and doing housework, as the disease progresses. Ultimately, pain and disability associated with the disease lead to a loss of functional independence and a profound reduction in quality-of- life. Impairments that are caused by KOA include knee pain, limited ROM of the knee, muscle weakness and knee instability.

The hip abductor muscles influence knee joint loading through their control of the pelvis in the frontal plane. Researchers have proposed that during the single-limb stance phase of gait, weakness of the stance-limb hip abductor muscles may lead to drop of the pelvis toward the contralateral limb, shifting the body's center of mass away from the stance limb toward the swing side. These adjustments, theoretically, could lead to higher knee adduction moments and greater medial knee joint loading.

Knee adduction moment is the moment that acts on the joint in the frontal plane. The knee adduction moment is generated by the combination of the ground reaction force, which passes medial to the centre of the knee joint during gait, and the perpendicular distance of this force from the centre of the joint. . This moment tends to adduct the tibiofemoral joint, causing an increase in medial compartment pressure, and people with knee OA have demonstrated larger than normal peak knee adduction moments in their gait patterns.

OA of the knee is characterized by changes in gait kinematics. High dynamic loads of the medial knee, as assessed by the external peak knee adduction moment, have been associated with tibiofemoral OA severity progression, and knee pain. The aging process impairs postural control more in a medial-lateral (ML) direction than in an anterior-posterior (AP) direction, which is linked with increased falling risk. Postural control stability in the ML direction, in orthostatic stance and during compensatory step, is dependent on hip abductor-adductor muscle torque .The hip abductor muscles are also needed to stabilize the lumbar-pelvic joint during gait and during balance recovery after external disturbance (postural responses of hip and step) This study aims to find the effect of hip abductor strengthening exercises on improving range of motion, functional activities, balance and minimizing pain in individuals affected by the knee OA.

ELIGIBILITY:
Inclusion Criteria:

* • Age group 40-60

  * Both genders male and female
  * Have had knee pain for 3 months or more
  * Report a minimum average overall pain severity of 4 on an 11-point numeric rating scale (NPRS) over the previous week
  * grade II and III on X-ray (Kellgren and Lawrence classification);
  * For participants with bilateral knee osteoarthritis, the more seriously affected side (as identified by the Kellgren-Lawrence grade of knee osteoarthritis and the pain intensity) was selected as the affected leg.
  * willing to participate in intervention program

Exclusion Criteria:

* • history of surgery of lower limb

  * Past knee fracture or malignancy
  * individuals with known hip OA and/or previous trauma affecting one or both hips
  * Intraarticular corticosteroid injection into the knee within previous 3 months.
  * Pregnancy

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-02-16 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 3 weeks
  The Numeric Pain Rating Scale (NPRS) is a segmented numeric version of the visual analog scale which is used to assess pain. It scores ranges from 0-10, 0 means No pain and 10 means Severe pain. Patient will be asked to verbally report the pain score
Western Ontario and McMaster Universities Osteoarthritis Index | 3 weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, validated questionnaire assessing pain, stiffness, and physical function in patients with knee osteoarthritis. It consists of 24 items divided into three subscales: Pain (5 items), Stiffness (2 items), and Physical Function (17 items).
Timed Up and Go test | 3 weeks
  The Timed Up and Go (TUG) test measures the time taken by a participant to stand up from a standard chair, walk a distance of 3 meters, turn around, walk back to the chair, and sit down. It assesses dynamic balance and functional performance.
Single leg stance | 3 weeks
  The Single leg stance (SLS) Test is used to assess static postural and balance control. Participants are instructed to stand on one leg unassisted, with eyes open and hands on hips. The duration for which the position is maintained is recorded.

SECONDARY OUTCOMES:
Range of Motion of Knee Joint | 3 weeks
  A goniometer will be used to measure the all the range of motion (ROM) of the knee joint

CONTACTS AND LOCATIONS:
Overall Officials: KINZA ANWAR, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- National Institute Of Rehabilitation Medicine G-8/2, Islamabad, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No